CLINICAL TRIAL: NCT04674930
Title: Effects of Home-based Exercise Program on Physical Functioning of Hemodialysis Patients.
Brief Title: Effects of Exercise Program on Physical Functioning of Hemodialysis Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/00703 Nahrat Kumar
Record Dates: First submitted 2020-12-16; First posted 2020-12-19 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Hemodialysis Patients
Keywords: Chronic kidney disease; Hemodialysis; Home-based exercise plan
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Pharmacological management
- Exercise group (Experimental): Aerobic training: The target training zone was set at 40-60% of the peak heart rate, as determined in the baseline 6min walk test (6MWT), with a rating of 11-13 on the Borg rating of perceived Exertion scale.
  Resistance Training: This training was prescribed at 70% of one repetition maximum (RM). Patients were instructed to train a variety of upper and lower body muscle groups (e.g., latissimus, deltoid, biceps, quadriceps, and gastrocnemius muscles), using Thera-band
  Interventions: Other: Exercise program

INTERVENTIONS:
Other: Exercise program — Home based exercise program including aerobic and resistance training will be carried out for a period of 6 weeks. Duration of aerobic exercise will be starting at 20 min/session, and progress to 30 ruin/session, with an increased pace according to the patient's capabilities. Resistance training with thera-band for 1 set of 10 repetitions twice a week. One RM will be reassessed weekly, and the program will be adjusted accordingly.
  Arms: Exercise group

SUMMARY:
This study is designed to provide a simple, home-based, low-moderate intensity exercise program in chronic renal disease patients who are undergoing hemodialysis in order to improve physical performance, decrease the level of fatigue and eventually increase quality of life in patients. A randomized control trial will be conducted including patients on hemodialysis, who will be randomly allocated to interventional and control groups. Both the groups will receive six weeks of treatment, 3 times per week. Data will be collected at baseline, 3rd week and 6th week. Outcome measures include assessment of physical functioning including six-minute walk test, standing balance, 4-metre gait speed, chair stand, fatigue assessment scale and quality of life in kidney disease patients on hemodialysis.

DETAILED DESCRIPTION:
Chronic Kidney Disease (CKD) is defined as the structural and functional abnormalities of kidney along with decreased Glomerular Filtration Rate (GFR) < 60 ml/min/1.73 m2 for 3 months. It also refers to an irreversible deterioration in renal function that usually develops over a period of years it represents not only as a biochemical abnormality but, eventually, loss of the excretory, metabolic and hormonal functions of the kidney which leads to the clinical symptoms and signs of renal failure. The alarmingly high prevalence of reduced GFR in adult men and women in Pakistan is not unexpected as the prevalence of risk factors of CKD including hypertension and diabetes is one of the highest reported worldwide. The prevalence rate of CKD is found to be 70% in Pakistan. Clinical sign of raised urea and creatinine should be found during routine blood tests. An early symptom is nocturia, tiredness or breathlessness, renal anemia or fluid overload, pruritus, anorexia, weight loss, nausea, vomiting and hiccups. In very advanced (chronic stage) renal failure, respiration may be particularly deep (Kussmaul breathing), metabolic acidosis, and patients may develop muscular twitching, fits, drowsiness and coma. Chronic kidney disease can be managed by lifestyle modifications (dietary management, weight management, physical activity) are the initial components of treatment. Blockade of the renin angiotensin aldosterone system, blood pressure control, optimally managed comorbid diabetes and avoidance of nephrotoxic medications to prevent worsening renal function are also part of management. Hemodialysis is a medical procedure to remove the waste products in the form of fluid from the blood and to correct electrolyte imbalances. This is accomplished using a machine and a dialyzer, also referred to as an artificial kidney. As dialysis requires patients to be seated for extended periods of time, the risk of developing obesity, high blood pressure, decreased quality of life, musculoskeletal problems, such as low back pain and muscle tightness is higher than normal.

The physiotherapeutic exercise program during hemodialysis improves the quality of life (QOL) of chronic renal patients in physical, social, environmental and psychological. On regular basis physiotherapy intervention is to a lower frequency of edema and muscle cramps and to reduce the intensity of pain. It also influences the improvement of the respiratory function, showed by the evolution of the values maximal inspiratory pressure (IPmax), maximal expiratory pressure (EPmax) and peak expiratory flow.

Studies reported that aerobic as well as strength training proved to have favorable short and long-term effects on the physical performance and the functional balance in patients on maintenance renal hemodialysis.

All patients undertaking hemodialysis (HD) are recommended to exercise to some extent. Intra-dialytic resistance training program is also feasible and effective, causing improvement in physical functioning by improving the strength, exercise capacity and performance in physical tests. Patients with chronic renal failure on hemodialysis, inspiratory muscle training induces improvement in respiratory muscle strength, functional capacity, lung function and quality of life. Inspiratory muscle training can improve maximal respiratory pressures, lung function, functional capacity and quality of life in patients with chronic renal failure who are receiving hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undertaking hemodialysis sessions for last 3 months
* Hemodynamically stable patients
* Stable clinical and functional state for at least 4 weeks
* Conscious level preserved
* Stage 5, Kidney Failure (GFR <15)

Exclusion Criteria:

* Patients with acute illness or infection, recent surgery, or vascular intervention
* Hospitalized within past 4 weeks (with dialysis or non-dialysis reasons)
* Uncontrolled Hypertension
* Patients with difficulty walking, without a walking aid owing to orthopedic problems
* Patients with neurological, musculoskeletal, cardiac and pulmonary disease and physical impairment

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Change in Six minute Walk test | 3 and 6 weeks of intervention
  This is a sub-maximal exercise test used to assess endurance and functional capacity. The distance covered in 6 minutes, is used as the outcome, by which we compare the changes in performance capacity. This test is performed in a gallery having a distance of 20m in length, in a straight line. In starting, the patient rests for 5 minutes in a sitting position, after 5 minutes the vitals will be assessed in resting phase. The patients are instructed about the test method, during one- minute intervals patients can ask about the time remaining during the test, prior to the end of the test. The distance walked in meters is then noted and functional capacity is estimated.

SECONDARY OUTCOMES:
Short Performance Physical Battery test (SPPB) | 3 and 6 weeks
  The SPPB examines three subcomponents of the lower extremity's function, these are standing balance, 4-metre gait speed, and chair stand these are of essential tasks for independent living among CKD patients on hemodialysis
Fatigue Assessment Scale (FAS) | 3 and 6 weeks
  Fatigue assessing scale can help in assessment of fatigue. The FAS is based on 10-item, which is used to evaluate symptoms of chronic fatigue. This is the self-reported questionnaire, measured by a notebook and pen, the time required to fulfill the self-assessment form is to take approximately 2 minutes
Kidney Disease Quality of Life - Short form (SF 36) (KDQOL-SF 36) | 3 and 6 weeks
  The KDQOL-36 is a self-administered to assess quality of life in patients with renal diseases. It requires paper- and-pencil and takes approximately 5 minutes to be filled. It assesses quality of life with regard to different domains of health

CONTACTS AND LOCATIONS:
Overall Officials: Suman Sheraz, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Rawalpindi, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] Gansevoort RT, Correa-Rotter R, Hemmelgarn BR, Jafar TH, Heerspink HJ, Mann JF, Matsushita K, Wen CP. Chronic kidney disease and cardiovascular risk: epidemiology, mechanisms, and prevention. Lancet. 2013 Jul 27;382(9889):339-52. doi: 10.1016/S0140-6736(13)60595-4. Epub 2013 May 31. PMID 23727170
- [Background] de Medeiros AIC, Fuzari HKB, Rattesa C, Brandao DC, de Melo Marinho PE. Inspiratory muscle training improves respiratory muscle strength, functional capacity and quality of life in patients with chronic kidney disease: a systematic review. J Physiother. 2017 Apr;63(2):76-83. doi: 10.1016/j.jphys.2017.02.016. Epub 2017 Mar 14. PMID 28433237
- [Background] Hall YN, Larive B, Painter P, Kaysen GA, Lindsay RM, Nissenson AR, Unruh ML, Rocco MV, Chertow GM; Frequent Hemodialysis Network Trial Group. Effects of six versus three times per week hemodialysis on physical performance, health, and functioning: Frequent Hemodialysis Network (FHN) randomized trials. Clin J Am Soc Nephrol. 2012 May;7(5):782-94. doi: 10.2215/CJN.10601011. Epub 2012 Mar 15. PMID 22422538
- [Background] Segura-Orti E, Kouidi E, Lison JF. Effect of resistance exercise during hemodialysis on physical function and quality of life: randomized controlled trial. Clin Nephrol. 2009 May;71(5):527-37. doi: 10.5414/cnp71527. PMID 19473613
- [Background] Davison SN, Tupala B, Wasylynuk BA, Siu V, Sinnarajah A, Triscott J. Recommendations for the Care of Patients Receiving Conservative Kidney Management: Focus on Management of CKD and Symptoms. Clin J Am Soc Nephrol. 2019 Apr 5;14(4):626-634. doi: 10.2215/CJN.10510917. Epub 2019 Feb 28. PMID 30819670
- [Background] Neto JR, Figueiredo E Castro LM, Santos de Oliveira F, Silva AM, Maria Dos Reis L, Quirino AP, Dragosavac D, Kosour C. Comparison between two physiotherapy protocols for patients with chronic kidney disease on dialysis. J Phys Ther Sci. 2016 May;28(5):1644-50. doi: 10.1589/jpts.28.1644. Epub 2016 May 31. PMID 27313390
- [Background] Uchiyama K, Washida N, Morimoto K, Muraoka K, Kasai T, Yamaki K, Miyashita K, Wakino S, Itoh H. Home-based Aerobic Exercise and Resistance Training in Peritoneal Dialysis Patients: A Randomized Controlled Trial. Sci Rep. 2019 Feb 22;9(1):2632. doi: 10.1038/s41598-019-39074-9. PMID 30796338